CLINICAL TRIAL: NCT05354778
Title: HYDROcortisone Versus Placebo for Severe HospItal-acquired Pneumonia in Intensive Care Patients: the HYDRO-SHIP Study
Acronym: HYDRO-SHIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo (Other)
Collaborators: Instituto do Cancer do Estado de São Paulo (Other); Hospital de Câncer de Barretos (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, João manoel Silva Junior, Principal Investigator, Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 54214821.0.1001.0068
Record Dates: First submitted 2022-04-20; First posted 2022-04-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Healthcare-Associated Pneumonia; Ventilator Associated Pneumonia
Keywords: Hydrocortisone; Intensive Care Unit; Pneumonia; Steroids; Critical Care
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated; Pneumonia | interventions — Hydrocortisone; hydrocortisone hemisuccinate

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, open-label clinical trial with two parallel groups: hydrocortisone and placebo. Data analyzed as "intention-to-treat".
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline 100mL every 8 hours for 5 days or until patient dies or is discharged from the intensive care unit
  Interventions: Drug: Placebo
- Hydrocortisone (Active Comparator): Hydrocortisone 100mg + normal saline 100mL every 8 hours for 5 days or until patient dies or is discharged from the intensive care unit
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Corticosteroid
  Other Names: Solu-CORTEF
  Arms: Hydrocortisone
Drug: Placebo — Normal saline only
  Other Names: NS
  Arms: Placebo

SUMMARY:
The use of corticosteroids in patients with severe community pneumonia, bacterial infection which kills lots of patients around the world, reduces the mortality of this infection. However, there are no studies with this type of drug regarding hospital-acquired pneumonia. This is the first multicenter randomized trial to test hydrocortisone plus standard therapy in critical care patients with nosocomial pneumonia. This intervention is inexpensive and may improve the outcome of those patients, besides having an acceptable side effects profile.

DETAILED DESCRIPTION:
Introduction and Objectives: the use of corticosteroids in patients with severe community pneumonia reduces morbimortality. However, to our knowledge, there are no studies with steroids for patients in intensive care with nosocomial pneumonia, among which those with ventilator associated pneumonia, infections which carry a high mortality rate. The treatment for those diseases involves intensive care and antibiotics, but there is a need for inexpensive, adjuvant therapies which improve the outcome for those patients. Therefore, the objective of this study is to compare hydrocortisone versus placebo, both with standard therapy, in the outcome of critical care patients diagnosed with nosocomial pneumonia. Methods: multicenter randomized, open-label, controlled trial, with two parallel groups: hydrocortisone or placebo, associated with nosocomial pneumonia's standard treatment. Patients with viral or other etiologies of pneumonia are excluded, as well as corticosteroids chronical users, or patients with conditions which demand this type of therapy. Intravenous 100mg of hydrocortisone and normal saline (the placebo) are tested every eight hours for five days or until intensive care unit (ICU) discharge or until the patient dies. The sample is 180 patients, 90 in each group, in different ICUs in Brazil. The primary outcome is early clinical failure. The secondary outcomes are survival and mortality in both groups, need for intubation, mechanical ventilation, vasoactive drugs and dialysis, lengths of stay in the hospital and in the ICU, radiological progression and adverse events. Discussion, risks, and benefits: this is the first multicenter randomized trial to test hydrocortisone plus standard therapy in critical care patients with nosocomial pneumonia. This intervention is inexpensive and may improve the outcome of those patients, besides having an acceptable side effects profile. Weighing the benefits and risks of this study, as well as its strengths and potential weaknesses, it is believed that its realization is justified, in addition to bringing important advances in the field of intensive care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Suspected ou confirmed case of bacterial nosocomial pneumonia (including ventilator-associated pneumonia)
* Intensive Care Unit stay
* Signed consent form (by the patient or a legal guardian)

Exclusion Criteria:

* Women who are pregnant, have recently given birth or are breastfeeding
* Patients who are moribund or do not have a treatment perspective
* Patients with community acquired pneumonia
* Patients with other types of pneumonia (viral - including COVID-19, fungal etc.)
* Those with pulmonary infiltrates in chest image which are not compatible with bacterial pneumonia
* Patients with adrenal insufficiency
* Patients who have a condition that demands the use of corticosteroids (acute or chronic)
* Patients allergic to hydrocortisone
* Patients with refractory septic shock (those receiving more than 0,5mcg/kg/min of norepinephrine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-10-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Early Clinical Failure | Between days 0 and 7 for death; between days 3 and 7 for respiratory or cardiovascular worsening
  Composite outcome: Death OR Respiratory worsening OR Cardiovascular worsening

SECONDARY OUTCOMES:
Survival | Days 7 and 28
  In the intensive care unit and in the hospital
Respiratory failure | 7 days
  Need for mechanical ventilation
Septic shock | 7 days
  Need for vasoactive drugs
Time of mechanical ventilation | 7 days
  Number of days patients require invasive ventilation support
Ventilator parameters (1) | 7 days
  Positive end expiratory pressure (PEEP)
Ventilator parameters (2) | 7 days
  Inspired oxygen fraction (FiO2)
Arterial blood gas analysis | 7 days
  Partial pressure of oxygen (PaO2)
Respiratory condition | 7 days
  Horowitz index for lung function (P/F ratio) - obtained from PaO2/FiO2
Time of vasoactive drugs use | 7 days
  Dosage and types of vasoactive drugs
Length of stay | 28 days
  In the Intensive Care Unit and in the hospital
Need for renal substitution therapy | 7 days
  Need for dialysis
Radiological worsening | 7 days
  Progression of image in the chest X-ray image
Adverse effects | 7 days
  psychosis, insomnia, hyperglycemia, hypernatremia, rhabdomyolysis, gastrointestinal bleeding and critical myopathy illness

CONTACTS AND LOCATIONS:
Overall Officials: João Manoel Silva Junior, MD, Principal Investigator — Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo
Locations (1):
- Hospital do Servidor Publico Estadual, São Paulo, Sao Paulo SP, Brazil

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Annane D, Sebille V, Charpentier C, Bollaert PE, Francois B, Korach JM, Capellier G, Cohen Y, Azoulay E, Troche G, Chaumet-Riffaud P, Bellissant E. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA. 2002 Aug 21;288(7):862-71. doi: 10.1001/jama.288.7.862. PMID 12186604
- [Background] Sprung CL, Annane D, Keh D, Moreno R, Singer M, Freivogel K, Weiss YG, Benbenishty J, Kalenka A, Forst H, Laterre PF, Reinhart K, Cuthbertson BH, Payen D, Briegel J; CORTICUS Study Group. Hydrocortisone therapy for patients with septic shock. N Engl J Med. 2008 Jan 10;358(2):111-24. doi: 10.1056/NEJMoa071366. PMID 18184957
- [Background] Annane D, Renault A, Brun-Buisson C, Megarbane B, Quenot JP, Siami S, Cariou A, Forceville X, Schwebel C, Martin C, Timsit JF, Misset B, Ali Benali M, Colin G, Souweine B, Asehnoune K, Mercier E, Chimot L, Charpentier C, Francois B, Boulain T, Petitpas F, Constantin JM, Dhonneur G, Baudin F, Combes A, Bohe J, Loriferne JF, Amathieu R, Cook F, Slama M, Leroy O, Capellier G, Dargent A, Hissem T, Maxime V, Bellissant E; CRICS-TRIGGERSEP Network. Hydrocortisone plus Fludrocortisone for Adults with Septic Shock. N Engl J Med. 2018 Mar 1;378(9):809-818. doi: 10.1056/NEJMoa1705716. PMID 29490185
- [Background] Annane D, Pastores SM, Rochwerg B, Arlt W, Balk RA, Beishuizen A, Briegel J, Carcillo J, Christ-Crain M, Cooper MS, Marik PE, Umberto Meduri G, Olsen KM, Rodgers SC, Russell JA, Van den Berghe G. Guidelines for the Diagnosis and Management of Critical Illness-Related Corticosteroid Insufficiency (CIRCI) in Critically Ill Patients (Part I): Society of Critical Care Medicine (SCCM) and European Society of Intensive Care Medicine (ESICM) 2017. Crit Care Med. 2017 Dec;45(12):2078-2088. doi: 10.1097/CCM.0000000000002737. PMID 28938253
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] WHO Rapid Evidence Appraisal for COVID-19 Therapies (REACT) Working Group; Sterne JAC, Murthy S, Diaz JV, Slutsky AS, Villar J, Angus DC, Annane D, Azevedo LCP, Berwanger O, Cavalcanti AB, Dequin PF, Du B, Emberson J, Fisher D, Giraudeau B, Gordon AC, Granholm A, Green C, Haynes R, Heming N, Higgins JPT, Horby P, Juni P, Landray MJ, Le Gouge A, Leclerc M, Lim WS, Machado FR, McArthur C, Meziani F, Moller MH, Perner A, Petersen MW, Savovic J, Tomazini B, Veiga VC, Webb S, Marshall JC. Association Between Administration of Systemic Corticosteroids and Mortality Among Critically Ill Patients With COVID-19: A Meta-analysis. JAMA. 2020 Oct 6;324(13):1330-1341. doi: 10.1001/jama.2020.17023. PMID 32876694
- [Background] Stern A, Skalsky K, Avni T, Carrara E, Leibovici L, Paul M. Corticosteroids for pneumonia. Cochrane Database Syst Rev. 2017 Dec 13;12(12):CD007720. doi: 10.1002/14651858.CD007720.pub3. PMID 29236286
- [Background] Blum CA, Nigro N, Briel M, Schuetz P, Ullmer E, Suter-Widmer I, Winzeler B, Bingisser R, Elsaesser H, Drozdov D, Arici B, Urwyler SA, Refardt J, Tarr P, Wirz S, Thomann R, Baumgartner C, Duplain H, Burki D, Zimmerli W, Rodondi N, Mueller B, Christ-Crain M. Adjunct prednisone therapy for patients with community-acquired pneumonia: a multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2015 Apr 18;385(9977):1511-8. doi: 10.1016/S0140-6736(14)62447-8. Epub 2015 Jan 19. PMID 25608756
- [Background] Confalonieri M, Urbino R, Potena A, Piattella M, Parigi P, Puccio G, Della Porta R, Giorgio C, Blasi F, Umberger R, Meduri GU. Hydrocortisone infusion for severe community-acquired pneumonia: a preliminary randomized study. Am J Respir Crit Care Med. 2005 Feb 1;171(3):242-8. doi: 10.1164/rccm.200406-808OC. Epub 2004 Nov 19. PMID 15557131
- [Background] Harris LK, Crannage AJ. Corticosteroids in Community-Acquired Pneumonia: A Review of Current Literature. J Pharm Technol. 2021 Jun;37(3):152-160. doi: 10.1177/8755122521995587. Epub 2021 Feb 22. PMID 34752553
- [Background] Fernandez-Serrano S, Dorca J, Garcia-Vidal C, Fernandez-Sabe N, Carratala J, Fernandez-Aguera A, Corominas M, Padrones S, Gudiol F, Manresa F. Effect of corticosteroids on the clinical course of community-acquired pneumonia: a randomized controlled trial. Crit Care. 2011 Mar 15;15(2):R96. doi: 10.1186/cc10103. PMID 21406101
- [Background] Meijvis SC, Hardeman H, Remmelts HH, Heijligenberg R, Rijkers GT, van Velzen-Blad H, Voorn GP, van de Garde EM, Endeman H, Grutters JC, Bos WJ, Biesma DH. Dexamethasone and length of hospital stay in patients with community-acquired pneumonia: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Jun 11;377(9782):2023-30. doi: 10.1016/S0140-6736(11)60607-7. Epub 2011 Jun 1. PMID 21636122
- [Background] Mikami K, Suzuki M, Kitagawa H, Kawakami M, Hirota N, Yamaguchi H, Narumoto O, Kichikawa Y, Kawai M, Tashimo H, Arai H, Horiuchi T, Sakamoto Y. Efficacy of corticosteroids in the treatment of community-acquired pneumonia requiring hospitalization. Lung. 2007 Sep-Oct;185(5):249-255. doi: 10.1007/s00408-007-9020-3. Epub 2007 Aug 21. PMID 17710485
- [Background] Snijders D, Daniels JM, de Graaff CS, van der Werf TS, Boersma WG. Efficacy of corticosteroids in community-acquired pneumonia: a randomized double-blinded clinical trial. Am J Respir Crit Care Med. 2010 May 1;181(9):975-82. doi: 10.1164/rccm.200905-0808OC. Epub 2010 Feb 4. PMID 20133929
- [Background] Torres A, Sibila O, Ferrer M, Polverino E, Menendez R, Mensa J, Gabarrus A, Sellares J, Restrepo MI, Anzueto A, Niederman MS, Agusti C. Effect of corticosteroids on treatment failure among hospitalized patients with severe community-acquired pneumonia and high inflammatory response: a randomized clinical trial. JAMA. 2015 Feb 17;313(7):677-86. doi: 10.1001/jama.2015.88. PMID 25688779
- [Background] Modi AR, Kovacs CS. Hospital-acquired and ventilator-associated pneumonia: Diagnosis, management, and prevention. Cleve Clin J Med. 2020 Oct 1;87(10):633-639. doi: 10.3949/ccjm.87a.19117. PMID 33004324
- [Background] Torres A, Niederman MS, Chastre J, Ewig S, Fernandez-Vandellos P, Hanberger H, Kollef M, Li Bassi G, Luna CM, Martin-Loeches I, Paiva JA, Read RC, Rigau D, Timsit JF, Welte T, Wunderink R. International ERS/ESICM/ESCMID/ALAT guidelines for the management of hospital-acquired pneumonia and ventilator-associated pneumonia: Guidelines for the management of hospital-acquired pneumonia (HAP)/ventilator-associated pneumonia (VAP) of the European Respiratory Society (ERS), European Society of Intensive Care Medicine (ESICM), European Society of Clinical Microbiology and Infectious Diseases (ESCMID) and Asociacion Latinoamericana del Torax (ALAT). Eur Respir J. 2017 Sep 10;50(3):1700582. doi: 10.1183/13993003.00582-2017. Print 2017 Sep. PMID 28890434
- [Background] Papazian L, Klompas M, Luyt CE. Ventilator-associated pneumonia in adults: a narrative review. Intensive Care Med. 2020 May;46(5):888-906. doi: 10.1007/s00134-020-05980-0. Epub 2020 Mar 10. PMID 32157357
- [Background] Metersky ML, Wang Y, Klompas M, Eckenrode S, Bakullari A, Eldridge N. Trend in Ventilator-Associated Pneumonia Rates Between 2005 and 2013. JAMA. 2016 Dec 13;316(22):2427-2429. doi: 10.1001/jama.2016.16226. No abstract available. PMID 27835709
- [Background] Dequin PF, Meziani F, Quenot JP, Kamel T, Ricard JD, Badie J, Reignier J, Heming N, Plantefeve G, Souweine B, Voiriot G, Colin G, Frat JP, Mira JP, Barbarot N, Francois B, Louis G, Gibot S, Guitton C, Giacardi C, Hraiech S, Vimeux S, L'Her E, Faure H, Herbrecht JE, Bouisse C, Joret A, Terzi N, Gacouin A, Quentin C, Jourdain M, Leclerc M, Coffre C, Bourgoin H, Lengelle C, Caille-Fenerol C, Giraudeau B, Le Gouge A; CRICS-TriGGERSep Network. Hydrocortisone in Severe Community-Acquired Pneumonia. N Engl J Med. 2023 May 25;388(21):1931-1941. doi: 10.1056/NEJMoa2215145. Epub 2023 Mar 21. PMID 36942789